CLINICAL TRIAL: NCT04282239
Title: Pectoral Nerves Block to Relieve Post-sternotomy Pain After Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not have the staff to conduct the study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01675
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Pain, Postoperative; Cardiac Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pectoral nerves block type 2 (PECS2) (Experimental): The intervention is the PECS2 block, a previously developed modality for preventing pain in the anterior chest. The medication used in the block is Ropivicaine 0.5%, Lidocaine 1% + 1:100,000 epinephrine, and 40 μg dexmedetomidine. Patients will receive a standard post-operative pain regimen per institutional protocol.
  Interventions: Procedure: PECS2 block; Drug: Ropivacaine 0.5% Injectable Solution; Drug: Lidocaine Epinephrine; Drug: Dexmedetomidine 0.004 MG/ML
- Control Group: standard post-operative pain regimen (No Intervention): Patients will receive a standard post-operative pain regimen per institutional protocol.

INTERVENTIONS:
Procedure: PECS2 block — Superficial peripheral nerve block placed at the interfascial plane between the pectoralis major and minor muscles and the plane between the pectoralis minor and serrates anterior muscles. Targeted nerves include the lateral and medial pectoral nerves in addition to the long thoracic nerve, thoracodorsal, and thoracic intercostal nerves from T2 to T6.
  Arms: Pectoral nerves block type 2 (PECS2)
Drug: Ropivacaine 0.5% Injectable Solution — 15 mL on each side of anterior chest for a total of 30mL
  Arms: Pectoral nerves block type 2 (PECS2)
Drug: Lidocaine Epinephrine — 10 mL on each side of anterior chest for a total of 20mL
  Arms: Pectoral nerves block type 2 (PECS2)
Drug: Dexmedetomidine 0.004 MG/ML — 10 mL
  Arms: Pectoral nerves block type 2 (PECS2)

SUMMARY:
The primary objective of this study is to determine if the addition of PECS2 block provides superior post-operative analgesia for cardiac surgery patients after midline sternotomy compared to only standard-of-care post-operative pain medication.

DETAILED DESCRIPTION:
The current study is a prospective, double-blind study investigating the use of pectoral nerves (PECS) block 2 to alleviate post-operative pain in cardiac surgery patients. The investigators anticipate enrolling a total of 220 participants in one of two groups, an interventional PECS block group and a control group not receiving the block. The intervention will occur in the operating room after the completion of the cardiac procedure and prior to the transfer of the participants to the cardiothoracic intensive care unit (CTICU). Both groups will receive the standard-of-care (SOC) pain regimen; the intervention with receive the PECS block in addition to SOC pain regimen. The procedure takes approximately five to ten minutes and will be conducted by the attending cardiac anesthesiologist. Pain will then be monitored hourly in the post-operative period in the CTICU. Additional measures will be investigated that are regularly logged in the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Obtaining one or more of the following elective surgical procedures at NYU Winthrop Hospital with midline sternotomy:

   * Coronary artery bypass graft (any number of vessels)
   * Aortic Valve Replacement (AVR)
   * Aortic Valve Repair
   * Mitral Valve Replacement (MVR)
   * Mitral Valve Repair
   * Tricuspid Valve Replacement
   * Tricuspid Valve Repair
   * Pulmonic Valve replacement
   * Pulmonic Valve Repair
   * Congenital Heart Defect Repair
   * Ascending Thoracic Aortic Aneurism Repair
   * Patient Age > 18 years.
2. Willingness and ability to participate in the study procedures
3. Sufficiently hemodynamically stable to give consent

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Hemodynamic instability
* Preexisting infection at site of block
* Allergy to block agents
* Severe psychiatric illness
* Intubated emergently prior to reception by the perioperative team
* Patient is preoperatively on extracorporeal membrane oxygenation (ECMO) treatment.
* Pregnant patient
* Recent surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Score on Critical-Care Pain Assessment Tool (CPOT) | 24 hours
  Measured at least hourly prior to extubation. This is an 8-item pain inventory seen as one of the top modalities for measuring pain in critical care patients. Minimum score of 0 and a maximum score of 8 (higher score = higher pain level).
Score on Visual Analog Scale (VAS) | 24 hours
  Measured at least hourly after extubation. 10 point pain analog scale (0-10, where 0 is no pain and 10 is highest pain level)

SECONDARY OUTCOMES:
Ventilatory duration post-operatively | 0-6 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is a time scale with the time of 0 corresponding to the "out of operating room" time and the final time being the time period from the 0 time to the time when the patient is extubated.
Duration of surgery | 4-6 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR (Electronic Medical Records). The scale is a time scale with the time of 0 corresponding to the "first incision" time and the final time being the time period from the 0 time to the time when the PECS2 block is completed.
Duration of operating room time | 5-7 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is a time scale with the time of 0 corresponding to the "into operating room" time and the final time being the "out of operating room" time
Total intraoperative fentanyl dose | Intraoperative duration
  Documented by anesthesia physician as standard of care - will be retrieved in the EMR.
  The scale is an absolute dosing scale in grams. It will be corrected for by weight (kilograms).
Duration of ICU stay | 24-48 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is time. Time zero is "out of operating" time and end time is time of downgrade or discharge from the hospital.
Duration of hospital stay | 5-7 days post-operative
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is a time with time zero corresponding to admission to hospital time and end time being the time of discharge from the hospital.
Time to first opiate dose for breakthrough pain | 24-48 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is time. Time zero will be "out of operating room" time and end time will be time of administration of first opiate pain medication.
Time to first analgesic post-operatively | 24-48 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is time. Time zero will be "out of operating room" time and end time will be time of administration of first breakthrough pain medication.
Number of episodes of post-operative breakthrough pain | 24-48 hours
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR. The scale is an absolute number documenting the number of documented episodes of breakthrough pain.
Total post-operative opiate dose | 5-7 days post-operative
  Documented by registered nurse as standard of care - will be retrieved in the EMR. The scale is an absolute dosing scale in grams. It will be corrected for by weight (kilograms).
Score on Critical-Care Pain Assessment Tool (CPOT) at 24-48h | 24-48 hours
  This is an 8-item pain inventory seen as one of the top modalities for measuring pain in critical care patients. Minimum score of 0 and a maximum score of 8 (higher score = higher pain level).
  Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR
Score on Visual Analog Scale (VAS) at 24-48h | 24-48 hours
  10 point pain analog scale (0-10, where 0 is no pain and 10 is highest pain level) Documented by nursing, physician assistants, physician, and/or respiratory staff as standard of care - will be retrieved in the EMR
Number of adverse events related to safety of the nerve block | 5-7 days post-operative
  Adverse events including but not limited to hemodynamic instability, respiratory depression, allergic reaction, shivering.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Abrol, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to sunil.abrol@nyulangone.org and harrison.pravder@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.